CLINICAL TRIAL: NCT02083692
Title: Pilot Study of Metformin in Head and Neck Squamous Cell Cancer and Its Effects on Stromal-epithelial Metabolic Uncoupling.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13D.458; JT 3153 (Other: JeffTrial Number)
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Cancer
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
The purpose of this study is to assess the effect of metformin in tumor metabolism in patients with head and neck cancer by evaluating metformin's ability to decrease TOMM20 expression in squamous carcinoma cells and decrease MCT4 expression in fibroblasts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck cancer biopsy proven, and who have a scheduled appointment for definitive resection of the tumor at TJUH
* Age ≥ 18 years of age and ≤80 years old.
* Newly diagnosed with HNSCC cancer.
* No prior therapy for HNSCC cancer is permitted for enrollment in the trial.
* All subjects must be able to comprehend and sign a written informed consent document.

Exclusion Criteria:

* Pregnant or may become pregnant during metformin administration.
* On metformin for any reason during the preceding 4 weeks.
* Diabetic patients are eligible if they are not taking metformin, insulin or sulfonylureas.
* Received iodinated contrast dye less than 48 hours prior to screening meet a temporary exclusion criteria to receive metformin. These patients cannot start investigational metformin until 48 hours have elapsed from contrast administration. Subjects who are scheduled for iodinated contrast dye administration within 48 hours of definitive surgery are excluded.
* Plasma alanine aminotransferase greater than 40 IU/dL.
* Plasma aspartate aminotransferase greater than 45 IU/dL.
* Plasma creatinine level greater than 1.3 mg/dL.
* Plasma alkaline phosphatase greater than 190 IU/dL.
* Plasma bicarbonate less than 22 mEq/L or history of lactic or any other metabolic acidosis.
* History of congestive heart failure.
* Myocardial ischemia or peripheral muscle ischemia.
* Sepsis or severe infection.
* History of lung disease currently requiring any pharmacologic or supplemental oxygen treatment.
* Scheduled for definitive HNSCC cancer surgical resection less than two weeks from enrollment or greater than five weeks from enrollment.
* History of hepatic dysfunction or hepatic disease.
* Excessive alcohol intake which is defined in accordance with CDC definitions as more than 1 drink per day for women and more than 2 drinks per day for men.

All medications are permitted except those that are contraindicated with metformin under current FDA recommendations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Change in TOMM20 and MCT4 expression from tumor cells from date of biopsy and date of surgery | date of biopsy and date of surgery (9-28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Curry, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Crist M, Yaniv B, Palackdharry S, Lehn MA, Medvedovic M, Stone T, Gulati S, Karivedu V, Borchers M, Fuhrman B, Crago A, Curry J, Martinez-Outschoorn U, Takiar V, Wise-Draper TM. Metformin increases natural killer cell functions in head and neck squamous cell carcinoma through CXCL1 inhibition. J Immunother Cancer. 2022 Nov;10(11):e005632. doi: 10.1136/jitc-2022-005632. PMID 36328378
- [Derived] Amin D, Richa T, Mollaee M, Zhan T, Tassone P, Johnson J, Luginbuhl A, Cognetti D, Martinez-Outschoorn U, Stapp R, Solomides C, Rodeck U, Curry J. Metformin Effects on FOXP3+ and CD8+ T Cell Infiltrates of Head and Neck Squamous Cell Carcinoma. Laryngoscope. 2020 Sep;130(9):E490-E498. doi: 10.1002/lary.28336. Epub 2019 Oct 8. PMID 31593308
- [Derived] Curry J, Johnson J, Tassone P, Vidal MD, Menezes DW, Sprandio J, Mollaee M, Cotzia P, Birbe R, Lin Z, Gill K, Duddy E, Zhan T, Leiby B, Reyzer M, Cognetti D, Luginbuhl A, Tuluc M, Martinez-Outschoorn U. Metformin effects on head and neck squamous carcinoma microenvironment: Window of opportunity trial. Laryngoscope. 2017 Aug;127(8):1808-1815. doi: 10.1002/lary.26489. Epub 2017 Feb 10. PMID 28185288
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/